CLINICAL TRIAL: NCT04138082
Title: Examining the Impact of Noise on Anesthesiologists' and Trainees' Situational Awareness in a High Fidelity Simulation Environment: a Prospective, Simulation-based, Randomized Trial
Brief Title: Impact of Noise on Anesthesiologists' and Trainees' Situational Awareness in a High Fidelity Simulation Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Jean-François Gagne, Anesthesiology Resident, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SituationalAwarenessNoise
Record Dates: First submitted 2019-10-16; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Noise; Adverse Effect
Keywords: Situational Awareness; Randomized-Control Trial; Medical Simulation; Patient Security

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blindly assigned to the high dB or low dB group. They were also blinded to the purpose of the study until completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dB Environment (Experimental): While performing the spinal anesthesia, the participants were exposed to a pre-recorded soundtrack of one of the investigators' operating rooms while the anesthesiology team was performing a spinal anesthesia. It included instruments noise and discussion but alarms, pulse oximetry and discussion with the patient were removed. The level of the soundtrack was set to be at 70 dB with peaks up to 100 dB, this level was recorded for every participant with Iphone™ application SoundMeter X 10.3 by Faber Acoustical, which has been both choosed in accordance with similar studies. The average noise was measured using the LEq value on a ''A'' scale (dB(A)) which correlate with frequencies perceived by the human ear. Speakers where placed at each corner of the room. Since literature describe that noise can initially enhance performance but is a transitory effect, the investigators decided to expose the experimental group to the maximum level of noise without any gradation.
  Interventions: Other: Exposition to high-dB soundtrack
- Low-dB Environment (No Intervention): The control group performed the same spinal anesthesia simulation scenario but without any soundtrack. The ambient noise in the room was recorded with the same method for each participant.

INTERVENTIONS:
Other: Exposition to high-dB soundtrack — Already stated
  Arms: High-dB Environment

SUMMARY:
The study is a single blinded randomized control trial. Participants were blinded to the purpose of the study and to the level of noise they would be exposed. Anesthesiology residents and certified anesthesiologists were recruited.The goal of this study was to measure the time needed to initiate treatment(TNIT) of a severe bradycardia while performing a spinal anesthesia in a high-fidelity simulation environment with either a low or a high ambient dB-level.

DETAILED DESCRIPTION:
Sample size To the investigators' knowledge, no similar study was done and predicting the difference in reaction time depending on level of noise is difficult. In comparable studies, sample size is small. The investigators then used a convenience sample based on the number of residents and staffs anesthesiologists who agreed to participate; the number of participants in this study exceeds the number of participants in previous research. Using the t value and the degrees-of-freedom of the unpaired t-test, the investigators calculated the effect size (r) to characterize the magnitude of the effect and evaluate if the sample size is enough to answer the research hypothesis. An r value of around 0.2 was considered a "weak" effect, 0.5 "medium", and 0.8 "strong". We recruited 15 participants in each group.

Simulation scenario The scenario was performed in situ in an operating room of the investigators' tertiary care hospital. It consisted of doing a spinal anesthesia for a 61 years old woman for a total hip replacement. She was known for stable asthma, high blood pressure and dyslipidemia. Upon entering the room, the anesthesiology evaluation and signed consentment were already completed. A simulated patient with a lumbar puncture simulator fixed on its back (Kyoto Kagaku M43B Lumbar Puncture Simulator II ®) was in position on the operating table for the technique. A simulated anesthesiology nurse was also present in the room. Standard monitoring with EKG, pulse oximeter, non invasive blood pressure were projected on a remotely controlled monitor with Castle Andersen ApS' SimMon app®. Simulated intravenous access was also already in place with the possibility to inject drugs if needed.

The participant then proceeded to the technique. Upon completion of local anesthesia, a mild auto-resolutive drop in heart rate from 85 to 65 without any other hemodynamic change. This benign change was used to try addressing hyper vigilance which is often happening in simulation scenarios. At the moment of dural puncture, a vasovagal event happened. It consisted of a standardised progressive diminution of the heart rate from 80 bpm to 30 bpm. After 10 seconds, blood pressure would fall to 70/40 with appropriate alarms at standard levels. The simulated patient did not tell its discomfort spontaneously but answered to questions if asked. After appropriate treatment, (putting the patient in dorsal position, administration of vasopressors or parasympatholytics) vital signs normalised in less than 30 seconds. The participant was then assigned to complete a questionnaire in another room.

Data Collection All participants were filmed for further revision. Demographics were gathered with a questionnaire. Collected datas were age, sex, resident or anesthesiologist status, number of years as a certified anesthesiologist or year of residency and if a hearing deficit was previously diagnosed. Participants also rated scenario realism on a 1 to 5 Likert scale.

Noise sensitivity was measured with Weinstein's Noise Sensitivity Scale, a 21-items validated questionnaire

After completion, collected datas were explained to the participants, questions were answered and if needed a more complete debriefing was made.

ELIGIBILITY:
Inclusion Criteria:

* To be a certified anesthesiologist or anesthesiology resident
* To have at least two months of anesthesiology exposure
* To consent to the study

Exclusion Criteria:

* To refuse to participate
* To have a hearing impairment diagnosis that affected anesthesiology practice.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Time To Initiate Treatment of a severe bradycardia (TNIT) | Through scenario completion, an average of 30 minutes
  The time to treatment of the vasovagal event was measured in seconds from the beginning of the bradycardia to the moment of appropriate treatment as previously defined(putting the simulated patient in dorsal position, administration of vasopressors or parasympatholytics). The investigators use this time as an indirect and pragmatic measure of participants' situational awareness without the need to regularly stop the scenario as a Situation Awareness Rating Technique (SAGAT) would need.

SECONDARY OUTCOMES:
Time to completed the task | Through scenario completion, an average of 30 minutes
  The time to realize the task which is from the beginning of the technique (landmark palpation) until cerebro-spinal fluid is obtained.
Swedish Occupational Fatigue Inventory (SOFI)Score | Through scenario completion, an average of 30 minutes
  The Swedish Occupational Fatigue Inventory is a 5 category questionnaire to assess occupational fatigue.(Lack of energy, physical exertion,physical discomfort,lack of motivation and sleepiness). Each category is declined in 4 adjectives that the participant has to rate on a scale from 0 to 6 (low agreement to high agreement). Results are reported for each category as the sum of each of its adjective from 0 to 24 (from low occupational fatigue to high occupational fatigue.
NASA Task Load Index (NASA-TLX) Score | Through scenario completion, an average of 30 minutes
  The participant has to rate each 6 category on a continous scale of 21 points as shown below.
  * Mental Demand From very low to very high
  * Physical Demand From very low to very high
  * Temporal demand From very low to very high
  * Performance From perfect to failure (This scale in interpreted in a reverse way)
  * Effort From very low to very high
  * Frustration From very low to very high The next step for the participant is to do a pairwise comparison of each category by selection the most contributive.
  Results are presented with transformation of the 21 points to a 100 points scale as a rating from 0 to 100 ( Low to high task load) By using pairwise comparison, a weighted global result is also presented with a score from 0 to 100 (Low to high task load)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Gagné, MD, Principal Investigator — Université de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katz JD. Noise in the operating room. Anesthesiology. 2014 Oct;121(4):894-8. doi: 10.1097/ALN.0000000000000319. No abstract available. PMID 24878496
- [Background] Murthy VS, Malhotra SK, Bala I, Raghunathan M. Detrimental effects of noise on anaesthetists. Can J Anaesth. 1995 Jul;42(7):608-11. doi: 10.1007/BF03011878. PMID 7553997
- [Background] Stevenson RA, Schlesinger JJ, Wallace MT. Effects of divided attention and operating room noise on perception of pulse oximeter pitch changes: a laboratory study. Anesthesiology. 2013 Feb;118(2):376-81. doi: 10.1097/ALN.0b013e31827d417b. PMID 23263015
- [Background] Kurmann A, Peter M, Tschan F, Muhlemann K, Candinas D, Beldi G. Adverse effect of noise in the operating theatre on surgical-site infection. Br J Surg. 2011 Jul;98(7):1021-5. doi: 10.1002/bjs.7496. PMID 21618484
- [Background] Broom MA, Capek AL, Carachi P, Akeroyd MA, Hilditch G. Critical phase distractions in anaesthesia and the sterile cockpit concept. Anaesthesia. 2011 Mar;66(3):175-9. doi: 10.1111/j.1365-2044.2011.06623.x. PMID 21320085
- [Background] Drzymalski DM, Ceruzzi J, Camann WR. Noise in the obstetric operating room. Int J Obstet Anesth. 2017 Feb;29:87-88. doi: 10.1016/j.ijoa.2016.10.008. Epub 2016 Oct 28. No abstract available. PMID 27884668
- [Background] Fritsch MH, Chacko CE, Patterson EB. Operating room sound level hazards for patients and physicians. Otol Neurotol. 2010 Jul;31(5):715-21. doi: 10.1097/MAO.0b013e3181d8d717. PMID 20431500
- [Background] Wang X, Zeng L, Li G, Xu M, Wei B, Li Y, Li N, Tao L, Zhang H, Guo X, Zhao Y. A cross-sectional study in a tertiary care hospital in China: noise or silence in the operating room. BMJ Open. 2017 Sep 18;7(9):e016316. doi: 10.1136/bmjopen-2017-016316. PMID 28928180
- [Background] Fitzgerald G, O'Donnell B. "In somno securitas" anaesthetists' noise exposure in Orthopaedic operating theatres. Ir Med J. 2012 Jul-Aug;105(7):239-41. PMID 23008884
- [Background] Wright MC, Taekman JM, Endsley MR. Objective measures of situation awareness in a simulated medical environment. Qual Saf Health Care. 2004 Oct;13 Suppl 1(Suppl 1):i65-71. doi: 10.1136/qhc.13.suppl_1.i65. PMID 15465958
- [Background] Schulz CM, Endsley MR, Kochs EF, Gelb AW, Wagner KJ. Situation awareness in anesthesia: concept and research. Anesthesiology. 2013 Mar;118(3):729-42. doi: 10.1097/ALN.0b013e318280a40f. PMID 23291626
- [Background] Enser M, Moriceau J, Abily J, Damm C, Occhiali E, Besnier E, Clavier T, Lefevre-Scelles A, Dureuil B, Compere V. Background noise lowers the performance of anaesthesiology residents' clinical reasoning when measured by script concordance: A randomised crossover volunteer study. Eur J Anaesthesiol. 2017 Jul;34(7):464-470. doi: 10.1097/EJA.0000000000000624. PMID 28394819
- [Background] McNeer RR, Bennett CL, Dudaryk R. Intraoperative Noise Increases Perceived Task Load and Fatigue in Anesthesiology Residents: A Simulation-Based Study. Anesth Analg. 2016 Feb;122(2):512-25. doi: 10.1213/ANE.0000000000001067. PMID 26797555
- [Background] Feuerbacher RL, Funk KH, Spight DH, Diggs BS, Hunter JG. Realistic distractions and interruptions that impair simulated surgical performance by novice surgeons. Arch Surg. 2012 Nov;147(11):1026-30. doi: 10.1001/archsurg.2012.1480. PMID 22801787